CLINICAL TRIAL: NCT04396613
Title: Assessment of Wound Closure Techniques in Primary Spine Surgery Using SPY Intra-operative Angiography
Brief Title: Wound Closure Techniques in Primary Spine Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Arjun S. Sebastian, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-011744
Record Dates: First submitted 2020-02-17; First posted 2020-05-20 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Spinal Injuries
MeSH Terms: conditions — Spinal Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Running Subcuticular Suture (Active Comparator)
  Interventions: Procedure: Closure technique
- Interrupted Vertical Mattress Suture (Active Comparator)
  Interventions: Procedure: Closure technique
- Staple Closure Techniques (Active Comparator)
  Interventions: Procedure: Closure technique

INTERVENTIONS:
Procedure: Closure technique — Randomized assignment to one of three known, effective closure techniques

SUMMARY:
The Researchers are trying to determine if there is a difference in blood flow around a wound site when comparing three different types of wound closure techniques.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Primary diagnosis of spinal stenosis
* Surgical indication for 1 or 2 level posterior spinal decompression or fusion

Exclusion Criteria:

* Pregnant or Breastfeeding
* Previous posterior spinal surgery
* Systemic corticosteroid use
* Long-term anticoagulation treatment
* Diagnosis of diabetes mellitus
* Diagnosis of peripheral arterial disease
* Current smoker
* Active infection of any kind or chronic infection with HIV, Hepatitis C, or Syphilis
* Iodine Allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Lowest perfusion - 10 Adjacent | Baseline
  Lowest perfusion score per 10 measurements taken along the wound closure as a percentage of perfusion at a standard location (5cm above incision).

SECONDARY OUTCOMES:
Lowest perfusion - 10 Alongside | At time of procedure
  Lowest perfusion score per 10 measurements taken along the wound closure
Average perfusion - 10 Alongside | At time of procedure
  Average perfusion score per 10 measurements taken along the wound closure
Average perfusion - 10 Adjacent | At time of procedure
  Average perfusion score per 10 measurements taken along the wound closure as a percentage of perfusion at a standard location (5cm above incision).
Lowest perfusion - 20 Adjacent | At time of procedure
  Lowest perfusion score per 20 measurements taken 1cm on either side of the wound closure as a percentage of perfusion at a standard location (5cm above incision)
Lowest perfusion - 20 Sides | At time of procedure
  Lowest perfusion score per 20 measurements taken 1cm on either side of the wound closure.
Average perfusion - 20 Sides | At time of procedure
  Average perfusion score per 20 measurements taken 1cm on either side of the wound closure.

CONTACTS AND LOCATIONS:
Overall Officials: Arjun Sebastian, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No